CLINICAL TRIAL: NCT03457922
Title: Evaluating a Personalized Trans-Diagnostic Group Therapy for Anxiety
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tali Manber Ball, PhD, Postdoctoral Scholar, Stanford University
Other Study IDs: 44584
Record Dates: First submitted 2018-01-29; First posted 2018-03-08 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Therapy: Patients in the Stanford Department of Psychiatry and Behavioral Sciences who are enrolling in a trans-diagnostic anxiety therapy group will be invited to participate in research on group processes and outcomes.

SUMMARY:
This study is examining the impact of a therapy group for all anxiety disorders provided by the Stanford Department of Psychiatry and Behavioral Sciences's Psychosocial Treatment Clinic on anxiety symptoms, impairment, and access to quality mental health care.

DETAILED DESCRIPTION:
Anxiety disorders are prevalent, impairing, and often precede other psychiatric and medical comorbidity (Kessler et al, 2005). Cognitive Behavior Therapy (CBT) and Acceptance and Commitment Therapy (ACT) are effective, evidence-based treatments for anxiety disorders that can be delivered in either a group or individual format (Deacon & Abramowitz, 2004; Arch et al 2012). Traditionally, group therapy has been delivered a single diagnosis at a time. This presents challenges to care delivery, however, because a sufficient number of patients with the same diagnosis and the same availability in their schedule must be assembled in order to start a group. Fortunately, CBT and ACT can be used to target key trans-diagnostic constructs such as excessive worry, avoidance, and fear of negative evaluation that may occur in many anxiety diagnoses. Indeed, emerging research suggests these constructs may be closer to the etiological dysfunction in anxiety disorders than the diagnoses themselves and may therefore be the best treatment targets (Craske, 2012). Because of this, there is now movement towards trans-diagnostic approaches that flexibly apply core principles of CBT and ACT to any anxiety disorder.

Group therapy is a cost-efficient and effective care delivery model that is also generally acceptable to patients with anxiety disorders. However, individual therapy is often preferred (Sharp et al, 2004), perhaps due to greater personalization of care relative to standard group therapy. To address this concern the investigators aim to use a pre-treatment assessment to develop a personalized plan for each patient entering a trans-diagnostic anxiety group.

In order to evaluate the effectiveness of this approach, patients enrolled in the group who consent to participate in research will complete assessments of anxiety and related symptoms, quality of life, and cognitive function before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Enrolled in a trans-diagnostic group therapy for anxiety disorders in the Stanford Psychiatry & Behavioral Sciences' Psychosocial Treatment Clinic.
* English fluency

Exclusion Criteria:

* Unable to provide informed consent
* Acute safety concerns (e.g., suicidality requiring a higher level of care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research study will be offered to all patients enrolling in a trans-diagnostic anxiety therapy group in the Stanford Department of Psychiatry & Behavioral Sciences. The purpose of this study is to evaluate the effect of this therapy group, so participants will be limited to those enrolling in the group as part of their clinical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale [OASIS] | 12 weeks
  Measures overall anxiety severity and anxiety-related impairment due to any anxiety disorder. Total scores are computed by summing scores from all 5 items. Total score ranges from 0 to 20, with higher scores indicating higher severity and impairment of anxiety symptoms. Reduction in OASIS scores therefore indicates better outcome.

SECONDARY OUTCOMES:
Sheehan Disability Scale [SDS] | 12 weeks
  Measures disability. Total scores are computed by summing scores from all 3 items. Total score ranges from 0 to 30, with higher scores indicating greater disability. Reduction in SDS scores therefore indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tali M Ball, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Department of Psychiatry & Behavioral Sciences, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No